CLINICAL TRIAL: NCT07111546
Title: An Open-label, Multicenter, Phase II Clinical Study to Evaluate the Efficacy and Safety of LBL-024 in Combination With Other Drugs for the Treatment of Patients With Advanced Solid Tumour[Substudy Number 02(BTC&HCC)]
Brief Title: A Clinical Trial of LBL-024 Combination Drug in Patients With Advanced Solid Tumours[Substudy 02(BTC&HCC)]
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBL-024-CN004_02(BTC & HCC)
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumour
MeSH Terms: interventions — Injections; durvalumab; Cisplatin; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LBL-024+Gemcitabine Hydrochloride+Cisplatin/Durvalumab+Gemcitabine Hydrochloride+Cisplatin (Experimental): Cohort 1：
  Subjects were treated with LBL-024 combined with gemcitabine and cisplatin
  or durvalumab combined with gemcitabine and cisplatin.
  Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Durvalumab Injection; Drug: Cisplatin Injection; Drug: Gemcitabine Hydrochloride for Injection
- LBL-024+Bevacizumab (Experimental): Cohort 2：
  Subjects were treated with LBL-024 combined with Bevacizumab.
  Intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Bevacizumab Injection

INTERVENTIONS:
Drug: LBL-024 for Injection — Intravenous infusion.
  Other Names: LBL-024
Drug: Durvalumab Injection — Intravenous infusion.
  Other Names: Durvalumab
  Arms: LBL-024+Gemcitabine Hydrochloride+Cisplatin/Durvalumab+Gemcitabine Hydrochloride+Cisplatin
Drug: Cisplatin Injection — Intravenous infusion.
  Other Names: Cisplatin
  Arms: LBL-024+Gemcitabine Hydrochloride+Cisplatin/Durvalumab+Gemcitabine Hydrochloride+Cisplatin
Drug: Gemcitabine Hydrochloride for Injection — Intravenous infusion.
  Other Names: Gemcitabine Hydrochloride
  Arms: LBL-024+Gemcitabine Hydrochloride+Cisplatin/Durvalumab+Gemcitabine Hydrochloride+Cisplatin
Drug: Bevacizumab Injection — Intravenous infusion.
  Other Names: Bevacizumab
  Arms: LBL-024+Bevacizumab

SUMMARY:
An open-label, multicenter, phase II clinical study to evaluate the efficacy and safety of LBL-024 in combination with other drugs for the treatment of patients with advanced solid tumour.

DETAILED DESCRIPTION:
This trial is an open-label, multicenter, phase II clinical study of LBL-024 in combination with other drugs for the treatment of patients with Advanced biliary tract cancer (BTC) and hepatocellular carcinoma (HCC), to evaluate the efficacy and safety of LBL-024 combination therapy.The trial included two cohorts.

Cohort 1: This cohort will have a safety run-in period,a small number of subjects will be enrolled to receive LBL-024 Combination Administration. After the subjects completed the 21-day safety observation, the sponsor and investigator jointly assessed the safety and tolerability of the combination drugs. If the safety and tolerability are good, the extension study of combination administration will be continued, the subjects will be continued to be enrolled, and the randomized, open, positive control trial design will be adopted. Eligible subjects will be randomized to either the LBL-024 treatment arm or the control arm.

Cohort 2: This cohort will have a safety run-in period, a small number of subjects will be enrolled to receive LBL-024 Combination Administration. After completing the 21-day safety observation, the safety and tolerability of the combination drugs will be assessed. The sponsor and investigator assessed the safety and tolerability of the combination drugs as good,and then the cohort will continue to enroll subjects.

The trial will enroll up to 172 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen, visit schedule, laboratory test, and other requirements of the protocol, and voluntarily enroll in the study and sign the written informed consent.
2. Age 18-75 years (inclusive of boundaries) at the time of signing informed consent form.
3. The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) is 0~1.
4. The expected survival time is at least 12 weeks.
5. According to the evaluation of RECIST 1.1 standard, the subjects enrolled have at least one measurable lesion.
6. There is adequate organ and bone marrow function,Conforms to laboratory test results.
7. Males with fertility and females of childbearing age are willing to take effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug.

Exclusion Criteria:

1. Participation in clinical studies of antineoplastic agents within 4 weeks before the first use of study drug,or Subject is expected to receive any other form of systemic or local anti-tumor therapy outside the protocol during the study.
2. Use of immunomodulatory drugs within 2 weeks before the first use of study drug,Including but not limited to thymopeptide, interleukins, interferon, etc.
3. Patients with active infection and currently requiring intravenous anti-infective therapy.
4. Patients with clinically uncontrollable pleural effusion, pericardial effusion, ascites, and those requiring repeated drainage or medical intervention.
5. The patient has a Medical history of immunodeficiency, including HIV antibody positive.
6. Women during pregnancy or lactation.
7. History of mental illness (interfering with understanding or giving informed consent), drug abuse, alcoholism or drug addiction.
8. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-12-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Objective Response Rate (complete response (CR) + partial response (PR)), as assessed by Response Evaluation Criteria in Solid Tumors (RECIST 1.1), refers to the percentage of study subjects who achieve a complete response or partial response.

SECONDARY OUTCOMES:
Disease Control Rate(DCR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Percentage of participants achieving CR and PR and stable disease (SD).
Duration of Response(DOR） | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The period from the participants first achieving CR or PR to disease progression.
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum drug concentration in plasma after administration.
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  After administration,Time to reach maximum drug concentration in plasma.
immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jian zhou, Principal Investigator — Shanghai Zhongshan Hospital
Locations (6):
- China (6):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital (SRRSH) Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No